CLINICAL TRIAL: NCT05182359
Title: Pragmatic Impact of Proteomic Risk Stratification in Diabetes Mellitus
Acronym: PORTRAIT-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: SomaLogic, Inc. (Industry)
Responsible Party: Principal Investigator, Ian J. Neeland, MD, Director, UH Center for Cardiovascular Prevention, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20211340
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVD-T2D Informed Medical Management (Informed) (Other): The SomaSignal Metabolic Factors test results will be provided in the Open Label Extension; results will not be provided to provider and participant until study conclusion.
  Interventions: Other: SomaSignal Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) Test and SomaSignal Metabolic Factors test
- Standard of Care (Uninformed) (Other): The SomaSignal Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) and Metabolic Factors test results will be provided in the Open Label Extension; results will not be provided to provider and participant until study conclusion.
  Interventions: Other: SomaSignal Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) Test and SomaSignal Metabolic Factors test

INTERVENTIONS:
Other: SomaSignal Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) Test and SomaSignal Metabolic Factors test — The SomaSignal Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) test is used to predict the four-year likelihood of myocardial infarction, stroke, hospitalization for heart failure or death. It will be provided to the participant's ordering provider.

SUMMARY:
Single-center, prospective, 2:1 randomized controlled parallel-group study, with an open label extension to evaluate SomaSignal Informed Medical Management (informed) versus Standard of Care (uninformed).

DETAILED DESCRIPTION:
Primary Aim: To determine whether risk stratification from SomaLogic's Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) test leads to riskconcordant changes in prescriptions and/or medical management in patients with diabetes.

Secondary Aims:

Secondary Aim 1: To evaluate the perspectives of healthcare providers on the impact of SomaLogic's Cardiovascular Risk in Type 2 Diabetes (CVD-T2D) test risk calculator in clinical practice.

Secondary Aim 2: To enable future health economic analyses of the impact of precision risk-stratified treatment.

Secondary Aim 3: In an open-label extension, to determine the impact of additional Metabolic Factor test results (beyond the SomaSignal Cardiovascular Risk in Type 2 Diabetes (CVD-T2D)) on medical management of the previously uninformed group at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care at a University Hospitals location
* Patients 40-89 year of age
* Diagnosis of Type 2 Diabetes Mellitus
* Eligible for but not currently prescribed a SGLT2i or GLP1RA per drug label. This includes a diagnosis of type 2 diabetes plus established atherosclerotic cardiovascular disease or high risk for atherosclerotic cardiovascular disease (including age ≥55 years with coronary, carotid, or lower-extremity atherosclerotic disease) or heart failure or chronic kidney disease with or without albuminuria.
* Patients that are able to provide consent

Exclusion Criteria:

* Intolerance or contraindication for use of both GLP1RA and SGLT2i
* Use of SGLT2i or GLP1RA within the 3 months prior to enrollment
* History of, an active, or untreated malignancy, in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years prior to, or are receiving or planning to receive therapy for cancer, at screening
* Patients that have Systemic Lupus Erythematous (SLE)
* End-stage renal disease
* Pregnancy (as determined by self-report)
* Inability to understand English (since must be able to understand risk report which is not translated by the manufacturer)

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The relation of prescription rates of cardioprotective medications (SGLT2i or GLP1 RA) to CVD-T2D test risk assessment in the Informed group vs. Uninformed group. | 12 weeks
  Medical record will be reviewed by the study team to evaluate changes in treatment strategy using the rate of new prescriptions for these medications.

SECONDARY OUTCOMES:
Survey of healthcare providers on the impact of SomaLogic's CVD-T2D calculator on patient care, medication prescription, and risk perception. | 12 weeks
  A survey will be obtained from the referring providers to assess perceived impact of the SomaLogic CVD-T2D test on risk.

OTHER OUTCOMES:
Cost effectiveness of the SomaLogic CVD-T2D test in the Informed vs. Uninformed groups. | 1 year
  Cost effectiveness of additional therapies measured by the incremental cost-effectiveness ratio utilizing the projected costs related to changes in prescription rates over the Quality Adjusted Life Years (QALYs), which reflects quality and quantity of life from cardiovascular event rate reductions estimated from the protein predicted risks. The incremental cost-effectiveness ratio is a way of investigating whether an intervention yields sufficient value to justify its cost. We will compare the Informed group to the Uninformed group, and find the difference in average cost, and differences in average effectiveness. The ratio is the incremental cost-effectiveness ratio (ICER). The recommended measure for effectiveness is Quality Adjusted Life Years (QALYs), which reflects quality and quantity of life.
The change in prescription rates of cardioprotective medications (SGLT2i or GLP1 RA) after revealing the CVD-T2D and Metabolic Factors test results at the end of the study in the Uninformed group. | 20 weeks
  Medical record will be reviewed by the study team to evaluate changes in treatment strategy using the rate of new prescriptions for these medications.
The change in prescription rates of cardioprotective medications (SGLT2i or GLP1 RA) after revealing the Metabolic Factors test results at the end of the study in the Informed group. | 20 weeks
  Medical record will be reviewed by the study team to evaluate changes in treatment strategy using the rate of new prescriptions for these medications.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Neeland, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05182359/Prot_SAP_000.pdf